CLINICAL TRIAL: NCT05356221
Title: BC112 Cross-sectional Evaluation of the Subjective Performance and Satisfaction With Ponto Sound Processors
Brief Title: Cross-sectional Evaluation of the Subjective Performance and Satisfaction With Ponto Sound Processors
Acronym: BC112
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BC112
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Unilateral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Ponto Users: Users that have been fitted with a Bone Anhcored Sound Processor, Ponto
  Interventions: Device: Ponto Sound processor

INTERVENTIONS:
Device: Ponto Sound processor — Bone Anchored Hearing solution fitted to compensate for the subjects hearing loss

SUMMARY:
The study is a non-interventional, observational, cross-sectional, study on users of Ponto sound processors. The purpose of this study is to evaluate subjectively assessed hearing performance and satisfaction with Oticon Medical's sound processors fitted with the Genie Medical fitting software.

DETAILED DESCRIPTION:
The study is a non-interventional, observational, cross-sectional, study on users of Ponto sound processors. The purpose of this study is to evaluate subjectively assessed hearing performance and satisfaction with Oticon Medical's sound processors fitted with the Genie Medical fitting software. Subjects fitted with one or two Ponto sound processors will be invited to participate in an online survey. The survey contains questions about the subjectively experienced performance and satisfaction of the device. The survey can be filled out on computer, tablet or mobile phone and should take the participants about 10 minutes to fill out.

ELIGIBILITY:
Inclusion Criteria:

Online consent form filled out Has been fitted with at least one Ponto Sound Processor

Exclusion Criteria:

No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Users fitted with a Ponto sound processor
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Philipsson, Study Director — Oticon Medical
Locations (1):
- Oticon Medical, Somerset, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ponto Users
Started | 170
Completed | 153
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Ponto Users
Number analyzed (Participants) | 170
Age, Customized [Count of Participants; unit: Participants]
  Age of participants: <18 years | 6
  Age of participants: 18-65 years | 65
  Age of participants: >65 years | 73
  Age of participants: Unknown | 26
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 75
  Female | 93
  Prefer not to answer | 1
  Unknown | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 170
Current usage of device [Count of Participants; unit: Participants] | 163
Uni- or bilateral use [Count of Participants; unit: Participants]
  Unilateral | 138
  Bilateral | 21
  Unknown | 11
Softband or abutment fitting [Count of Participants; unit: Participants]
  Softband | 3
  Abutment | 156
  Unknown | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall IOI-HA Score
Description: International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1) to best outcome (5). Evaluate subjectively assessed overall hearing performance and satisfaction with the Oticon Medical's Ponto sound processors.
Time Frame: at enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ponto, Ponto Pro, & Ponto Plus; Ponto 3 & Ponto 3 Power; Ponto 3 SuperPower; Ponto 4; Ponto 5 Mini; Ponto 5 SuperPower: Type/model of Ponto sound processor
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
score on a scale | 3.98 (0.12) | 3.96 (0.12) | 3.86 (0.15) | 4.02 (0.15) | 4.22 (0.21) | 4.11 (0.12)

2. Secondary Outcome: Factor 1 IOI-HA Score
Description: Factor 1 International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1) to best outcome (5). Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollement
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
score on a scale | 4.2 (0.1) | 4.2 (0.1) | 4.1 (0.1) | 4.3 (0.1) | 4.6 (0.2) | 4.3 (0.1)

3. Secondary Outcome: Factor 2 IOI-HA Score
Description: Factor 2 International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1) to best outcome (5). Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
score on a scale | 3.7 (0.1) | 3.7 (0.1) | 3.5 (0.1) | 3.7 (0.2) | 3.8 (0.2) | 3.7 (0.1)

4. Secondary Outcome: Per Item IOI-HA Score (Q1)
Description: Per item International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1) to best outcome (5). Here, this item queries average hours of use per day and a score of 1 is assigned for "none", a score of 2 assigned for "less than one hour per day", a score of 3 assigned for "1 to 4 hours per day", a score of 4 for "4 to 8 hours a day", and a score of 5 assigned for "more than 8 hours a day". Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants
  None | 1 | 0 | 0 | 0 | 0 | 0
  Less than one hour a day | 2 | 3 | 1 | 1 | 0 | 1
  1 to 4 hours a day | 2 | 2 | 3 | 4 | 0 | 2
  4 to 8 hours a day | 7 | 2 | 3 | 6 | 1 | 5
  More than 8 hours a day | 30 | 13 | 12 | 31 | 8 | 13

5. Secondary Outcome: Per Item IOI-HA Score (Q2)
Description: Per item International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1: helped not at all) to best outcome (5: helped very much). Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants
  Helped not at all | 2 | 0 | 0 | 0 | 0 | 0
  Helped slightly | 3 | 1 | 0 | 5 | 0 | 1
  Helped moderately | 9 | 4 | 7 | 4 | 1 | 4
  helped quite a lot | 9 | 7 | 4 | 17 | 4 | 6
  Helped very much | 19 | 8 | 8 | 16 | 4 | 10

6. Secondary Outcome: Per Item IOI-HA Score (Q3)
Description: Per item International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1: Very much difficulty) to best outcome (5: No difficulty). Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants
  Very much difficulty | 1 | 1 | 1 | 3 | 0 | 1
  Quite a lot of difficulty | 3 | 3 | 1 | 1 | 3 | 2
  Moderate difficulty | 12 | 4 | 11 | 15 | 0 | 3
  Slight difficulty | 22 | 10 | 3 | 21 | 5 | 11
  No difficulty | 4 | 2 | 3 | 2 | 1 | 4

7. Secondary Outcome: Per Item IOI-HA Score (Q4)
Description: Per item International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1: Not worth it at all) to best outcome (5: Very much worth it). Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants
  Not at all worth it | 1 | 1 | 0 | 0 | 0 | 0
  Slightly worth it | 3 | 0 | 0 | 4 | 0 | 1
  Moderately worth it | 6 | 2 | 5 | 5 | 0 | 3
  Quite a lot of worth it | 7 | 5 | 4 | 7 | 2 | 3
  Very much worth it | 25 | 12 | 10 | 26 | 7 | 14

8. Secondary Outcome: Per Item IOI-HA Score (Q5)
Description: Per item International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1: Affected very much) to best outcome (5: Affected not at all). Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants
  Affected very much | 2 | 0 | 1 | 3 | 0 | 2
  Affected quite a lot | 4 | 2 | 3 | 4 | 1 | 1
  Affected moderately | 7 | 7 | 4 | 7 | 3 | 4
  Affected slightly | 20 | 7 | 7 | 20 | 4 | 9
  Affected not at all | 8 | 4 | 4 | 8 | 1 | 4
  Missing | 1 | 0 | 0 | 0 | 0 | 1

9. Secondary Outcome: Per Item IOI-HA Score (Q6)
Description: Per item International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1: bothered very much) to best outcome (5: Bothered not at all). Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants
  Bothered very much | 1 | 0 | 2 | 1 | 0 | 0
  Bothered quite a lot | 5 | 1 | 2 | 4 | 0 | 2
  Bothered moderately | 9 | 6 | 1 | 6 | 3 | 4
  Bothered slightly | 11 | 8 | 9 | 16 | 1 | 4
  Bothered not at all | 16 | 5 | 5 | 15 | 5 | 11

10. Secondary Outcome: Per Item IOI-HA Score (Q7)
Description: Per item International Outcome Inventory for Hearing Aids score. 5 item categorical scale ranging from worst outcome (1: Worse) to best outcome (5: Very much better). Evaluate the subjectively assessed performance and satisfaction with Oticon Medical's Ponto sound processors
Time Frame: at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants
  Worse | 0 | 1 | 0 | 0 | 0 | 0
  No change | 4 | 1 | 2 | 3 | 0 | 1
  Slightly better | 7 | 2 | 5 | 8 | 2 | 4
  Quite a lot better | 14 | 8 | 6 | 10 | 2 | 5
  Very much better | 17 | 8 | 6 | 21 | 5 | 11

11. Secondary Outcome: Usage
Description: Evaluate non-usage among patients fitted with a Ponto sound processor. Reported is number of participants by sound processor type.
Time Frame: at enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Upgrade
Description: Evaluate Ponto sound processor upgrade rate
Time Frame: enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
Number analyzed (Participants) | 42 | 20 | 19 | 42 | 9 | 21
Participants
  Yes | 16 | 11 | 12 | 23 | 5 | 12
  No | 25 | 9 | 7 | 19 | 4 | 9
  Did not answer | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Collection of adverse events not applicable since study is a non-interventional, observational, cross-sectional, survey investigation
Description: Collection of adverse events not applicable since study is a non-interventional, observational, cross-sectional, survey investigation
Arm/Group | Ponto, Ponto Pro, & Ponto Plus | Ponto 3 & Ponto 3 Power | Ponto 3 SuperPower | Ponto 4 | Ponto 5 Mini | Ponto 5 SuperPower
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Survey study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT05356221/Prot_SAP_000.pdf